CLINICAL TRIAL: NCT06293131
Title: Median Effective Dose of Ciprofol-Assisted Sedation for Elderly Patients Undergoing Knee Arthroplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, Professor, Second Hospital of Shanxi Medical University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: yuewei20230705
Record Dates: First submitted 2024-01-23; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Sedation; ED50; Knee Arthroplasty
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ciprofol-assisted sedation 1 (Experimental): Adjusting the dose of ciprofol-assisted sedation in knee arthroplasty on a case-by-case basis
  Interventions: Drug: Ciprofol

INTERVENTIONS:
Drug: Ciprofol — Ciprofol was injected intravenously, and was pumped during operation to maintain sedation
  Other Names: Ropivacaine

SUMMARY:
Regional anesthesia is a common clinical anesthesia method, and regional anesthesia-assisted sedation play a central role in promoting patient comfort and relieving anxiety. With increasing age, elderly people experience changes in pharmacokinetics and pharmacodynamics and increased drug sensitivity. Ciprofol has advantages in adverse events such as hypotension and respiratory depression. There are fewer studies on the recommended dosage of ciprofol-assisted sedation for intrathecal anesthesia in elderly patients. The aim of study is to identify the median effective dose(ED50) of ciprofol-assisted sedation in elderly patients undergoing spinal anesthesia

DETAILED DESCRIPTION:
Select the patients who received knee arthroplasty in the Second Hospital of Shanxi Medical University. The patients received a loading dosage of 0.05mg/kg of ciprofol to begin sedation following the completion of intravertebral anesthesia, and the maintenance dose is calculated using the sequential method. Based on the relevant literature and pilot study, 0.2 mg·kg-1·h-1 is selected as initial test dose with a dose gradient of 0.02 mg·kg-1·h-1. The Modified Alertness Sedation Score (MOAA/S ) scores and the bispectral index (BIS) were recorded for patients before administration (T0), 5 min after administration (T1), 10 min after administration (T2), 20 min after administration (T3), 30 min after administration (T4), 45 min after administration (T5), and 60min after administration (T6). If the first patient had ≥ 4 time points with MOAA/A score ≤3 and BIS<85 from T0-T6, the sedation was regarded as satisfactory, then the next patient 's dose of ciprofol was reduced by one level. On the contrary, if the patient's MOAA/S score and BIS at T0-T6 had less than 4 points of MOAA/S ≤3 points and BIS <85, it was regarded as unsatisfactory sedation. The next patient's dose of ciprofol was increased by one level. After 8 crossovers, the trial was terminated. At the same time, the change of vital signs and adverse reactions before and after administration were recorded

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* ASA grade I~III
* BMI 18~30 kg/m2

Exclusion Criteria:

* Contraindications to intrathecal anesthesia
* Suffering from severe psychiatric or neurologic disorders or taking sedative drugs within the last 3 months
* Difficult airway or having respiratory diseases such as upper airway obstruction
* Severe cardiovascular system diseases
* Severe hepatic or renal dysfunction
* Allergy or contraindication to propofol and its drug-related components
* Patient Prefusal

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Modified Alertness Sedation Score (MOAA/S) | 24 hours
  Changes in Modified Alertness Sedation Score
Bispectral index (BIS) | 24 hours
  Changes in Bispectral index

SECONDARY OUTCOMES:
systolic blood pressure （SBP） | 24 hours
  Changes in systolic blood pressure
diastolic blood pressure（DBP） | 24 hours
  Changes in diastolic blood pressure
heart rate (HR) | 24 hours
  changes in heart rate
pulse oxygen saturation（SpO2） | 24 hours
  changes in pulse oxygen saturation

OTHER OUTCOMES:
Occurrence of Sedation-related adverse events | 72 hours
  It includes intraoperative and postoperative sedation-related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China